CLINICAL TRIAL: NCT01332409
Title: Special Drug Use Investigation for ADOAIR DISKUS COPD (Salmeterol and Fluticasone)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113095
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients prescribed salmeterol and fluticasone: Patients with chronic obstructive pulmonary disease prescribed salmeterol and fluticasone during study period
  Interventions: Drug: Salmeterol and Fluticasone

INTERVENTIONS:
Drug: Salmeterol and Fluticasone — Administered according to the prescribing information in the locally approved label by the authorities.

SUMMARY:
To investigate possible problems or questions in safety and effectiveness of salmeterol and fluticasone in patients with chronic obstructive pulmonary disease (bronchitis chronic / emphysema). In this special drug use investigation, onset of pneumonia shall be handled as the priority investigation item.

ELIGIBILITY:
Inclusion Criteria:

* Must use salmeterol and fluticasone for the first time

Exclusion Criteria:

* Patients with hypersensitivity to salmeterol and fluticasone
* Patients with infection which salmeterol and fluticasone is not effective
* Patients with deep mycosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are diagnosed as having a chronic obstructive pulmonary disease (bronchitis chronic / emphysema)
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2009-08; Primary Completion 2012-04 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events in Japanese patients treated with salmeterol and fluticasone based on prescribing information under the conditions of general clinical practice. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Chiba, Japan

REFERENCES:
- [Background] Yoriko Morioka, Hiroharu Abe, Terufumi Hara, Pascal Yoshida. Post-marketing Surveillance of Salmeterol Xinafoate / Fluticasone Propionate (Adoair®250Diskus®) - Interim Report -. Resp Med - Kokyuki Naika. 2013;23(1):111-122.